CLINICAL TRIAL: NCT06097546
Title: Evaluation of Serum Retinoic Acid Induced Protein 14 (RAI14) and Metastasis Associated Cancer Colon -1 (MACC-1) as Biomarkers for Breast Cancer
Brief Title: Serum Retinoic Acid Induced Protein 14 (RAI14) and Metastasis Associated Cancer Colon -1 (MACC-1) in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Atef Mohamed Elbadry, Prinicipal investigator (doctor), Assiut University
Other Study IDs: Markers in Breast Cancer
Record Dates: First submitted 2023-10-07; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer patients: Newly diagnosed patients with breast cancer
  Interventions: Diagnostic Test: laboratory test (RAI14 and MACC-1 )
- Benign lesions: Diagnosed patients with benign breast lesions
  Interventions: Diagnostic Test: laboratory test (RAI14 and MACC-1 )
- Control: apparently healthy individuals with matched age and sex
  Interventions: Diagnostic Test: laboratory test (RAI14 and MACC-1 )

INTERVENTIONS:
Diagnostic Test: laboratory test (RAI14 and MACC-1 ) — Measurement of serum RAI14 and serum MACC-1 levels by immunochemical assays

SUMMARY:
1. Measurement of serum levels of Retinoic acid induced 14 (RAI14) and Metastasis associated cancer colon -1 (MACC-1) as biomarkers for diagnosis of breast cancer.
2. Study their relationship to disease stages and clinicopathological features of BC.
3. Compare the diagnostic performance of serum RAI14 and serum MACC-1 with serum Carcinoembryonic antigen (CEA) and Cancer antigen 15-3 (CA15-3) for diagnosis of BC.

DETAILED DESCRIPTION:
Breast cancer (BC) is one of the most prevalent Neoplasms and the second leading reason of death from cancer in women. Every year approximately 2.3 million new cases of BC are diagnosed worldwide. Due to the high impact of this type of cancer, the early detection, early diagnosis and effective treatment, will improve the diagnosis of patients and lower the associated mortality rates. Carcinoembryonic antigen (CEA) and Cancer antigen 15-3 (CA15-3) are the most commonly used serum markers in the diagnosis and follow up of BC, However their clinical applications still remain controversial.

Retinoic acid induced protein 14 (RAI14) is an actin-binding protein which participates in physiological processes such as the regulation of cell polarity and transport of spermatozoa. Recent studies showed that RAI14 is overexpressed in several malignant tumors with a significant role in the development of tumors . The serum RAI14 is a reliable novel marker in the early diagnosis and chemotherapy monitoring of triple-negative BC.

Metastasis-associated colon cancer-1 (MACC-1) is a newly identified tumor marker, first identified in colon cancer tissue as a prognostic indicator and inducer of metastasis .It is located on human chromosome 7 (7p21.1) and shown to be a key regulator of the hepatocyte growth factor-mesenchymal epithelial transition factor( HGF-MET) pathway in colon cancer. It is shown that serum MACC-1 can be a potential biomarker for diagnosis and progression in patients with BC. There was a strong correlation between MACC-1 expression and the clinical and the primary tumor, regional nodes, metastasis (TNM) stages of BC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with benign breast lesions.
2. Patients with breast cancer who were confirmed by histopathological studies and did not receive any treatment.

Exclusion Criteria: 1- Patients who received chemotherapy or radiotherapy. 2- Patients with known other organ malignancy.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study will be carried out on 3 groups
  * Group (1)(patient group):
    30 newly diagnosed patients with breast cancer, who will be admitted Clinical Pathology Department, Assiut University Hospitals, Assiut University Patients group will be furtherly subclassified according to the TNM staging classification .
  * Group (2) (benign lesions) 30 diagnosed patients with benign breast lesions.
  * Group (3) (control group):
    30 apparently healthy individuals with matched age and sex are included in this study as a control group for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic value of serum Retinoic acid induced 14 (RAI14) and Metastasis associated cancer colon -1 (MACC-1) for breast cancer patients. | Baseline
  Evaluation of the clinical utility of measurement of level of Retinoic acid induced 14 (RAI14) and Metastasis associated cancer colon -1 (MACC-1) in newly diagnosed breast cancer patients

SECONDARY OUTCOMES:
Correlate the levels of serum Retinoic acid induced 14 (RAI14) and Metastasis associated cancer colon -1 (MACC-1) with the TNM staging in breast cancer patients. | Baseline
  Studying the correlation of levels of serum Retinoic acid induced 14 (RAI14) and Metastasis associated cancer colon -1 (MACC-1) with the TNM staging in breast cancer patient.

REFERENCES:
- [Background] Cui R, Zou J, Zhao Y, Zhao T, Ren L, Li Y. The dual-crosslinked prospective values of RAI14 for the diagnosis and chemosurveillance in triple negative breast cancer. Ann Med. 2023 Dec;55(1):820-836. doi: 10.1080/07853890.2023.2177722. PMID 36880986
- [Background] Lv M, Jiao Y, Yang B, Ye M, Di W, Su W, Zhong J. MACC1 as a Potential Target for the Treatment and Prevention of Breast Cancer. Biology (Basel). 2023 Mar 16;12(3):455. doi: 10.3390/biology12030455. PMID 36979146
- [Background] Ahmed M, Aslam M. Serum MACC-1: a new biomarker for breast cancer. Oncotarget. 2020 Dec 1;11(48):4521-4526. doi: 10.18632/oncotarget.27813. eCollection 2020 Dec 1. PMID 33400729